CLINICAL TRIAL: NCT05856721
Title: Pattern of Intestinal Parasitic Infection Among Cirrhotic Patients in Sohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nada Nady Abdelaal, residant at Tropical Medicine & Gastroenterology departmrnt sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-23-04-13MS
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Occult Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases group (Active Comparator): One hundred patients with liver cirrhosis and GIT complaints
  Interventions: Diagnostic Test: stool analysis
- control group (Active Comparator): One hundred patients with GIT complaints but not have any cormobidity
  Interventions: Diagnostic Test: stool analysis

INTERVENTIONS:
Diagnostic Test: stool analysis — Detection of prevalence and pattern of intestinal parasitic infection in cirrhotic patients and the difference between cirrhotic patients and non-cirrhotic patients with no comorbidity.
  To determine the most common risk factors of intestinal parasitic infection in cirrhotic patients.

SUMMARY:
Chronic hepatic illness is one of the most serious health issues . Liver cirrhosis as the latest phase of chronic liver disease causes a disorder called cirrhosis-associated immune dysfunction syndrome (CAIDS) . Cirrhosis comes to be a systemic disease, with several organ disorders. At this phase, patients become highly vulnerable to various infections because of CAIDS, which comprises both innate and adaptive immunity). Patients with hepatic cirrhosis and ascites are more liable to other complications of liver disease, including hyponatremia, refractory ascites, or hepatorenal syndrome (HRS) . Liver cirrhotic patients are considered to be as immunosuppressed and are vulnerable to a different species of entero-parasites .

Intestinal parasitic diseases have been reported in association with diabetes mellitus (DM) which is considered a predisposing factor to infection in cirrhotic patients . Immunosuppression among DM cases is due to increased blood glucose levels, which modifies several immune responses and this renders the body susceptible to various opportunistic infections comprising parasitic infections

Intestinal parasites such as Blastocystis hominis, Cryptosporidium spp., Isospora belli, Cyclospora cayetanensis, and Microsporidia have appeared as significant opportunistic parasites that are responsible for severe illness in immunocompromised patients , subsequently, patients suffer from severe morbidity and high mortality).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have liver cirrhosis with or without hepatocellular carcinoma.

Exclusion Criteria:

* . Cirrhotic patients with renal impairment.
* . Cirrhotic patients with cardiac diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pattern of Intestinal Parasitic Infection Among Cirrhotic Patients | 12 months
  Detection of prevalence and pattern of intestinal parasitic infection in cirrhotic patients and the difference between cirrhotic patients and non-cirrhotic patients with no comorbidity.
  To determine the most common risk factors of intestinal parasitic infection in cirrhotic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arvaniti V, D'Amico G, Fede G, Manousou P, Tsochatzis E, Pleguezuelo M, Burroughs AK. Infections in patients with cirrhosis increase mortality four-fold and should be used in determining prognosis. Gastroenterology. 2010 Oct;139(4):1246-56, 1256.e1-5. doi: 10.1053/j.gastro.2010.06.019. Epub 2010 Jun 14. PMID 20558165
- [Background] Bernardi M, Moreau R, Angeli P, Schnabl B, Arroyo V. Mechanisms of decompensation and organ failure in cirrhosis: From peripheral arterial vasodilation to systemic inflammation hypothesis. J Hepatol. 2015 Nov;63(5):1272-84. doi: 10.1016/j.jhep.2015.07.004. Epub 2015 Jul 17. PMID 26192220
- [Background] Bonnel AR, Bunchorntavakul C, Reddy KR. Immune dysfunction and infections in patients with cirrhosis. Clin Gastroenterol Hepatol. 2011 Sep;9(9):727-38. doi: 10.1016/j.cgh.2011.02.031. Epub 2011 Mar 11. PMID 21397731
- [Background] El-Shazly LB, El-Faramawy AA, El-Sayed NM, Ismail KA, Fouad SM. Intestinal parasitic infection among Egyptian children with chronic liver diseases. J Parasit Dis. 2015 Mar;39(1):7-12. doi: 10.1007/s12639-013-0346-x. Epub 2013 Sep 3. PMID 25698851